CLINICAL TRIAL: NCT07402304
Title: The Cultivation of College Students' Social Behavior in Public Physical Education Courses in Colleges and Universities: A Study Based on the Experiential Learning Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Han Xu (Other)
Responsible Party: Sponsor-Investigator, Han Xu, Graduate Student, Yangzhou University
Organization: Yangzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: YXYLL -2025- 120
Record Dates: First submitted 2026-02-02; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Prosocial Behavior; Physical Literacy
MeSH Terms: conditions — Altruism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group: Tennis Course Based on Experiential Learning Model (Experimental): The experimental group will participate in a tennis course based on the experiential learning model. The course will involve 90-minute weekly sessions, focusing on tennis skill development and social interaction activities designed to promote cooperation and enhance prosocial behavior among students. This intervention aims to foster teamwork, social responsibility, and collective spirit through sports.
  Interventions: Behavioral: experiential learning model
- Control Group: Regular Tennis Course (Active Comparator): The control group will continue with the regular tennis course, focusing solely on tennis skill development without incorporating the experiential learning model. The course will follow the standard physical education curriculum without additional social interaction activities aimed at enhancing prosocial behavior or cooperation.
  Interventions: Behavioral: Regular Tennis Course

INTERVENTIONS:
Behavioral: experiential learning model — The intervention in this study consists of a tennis course based on the experiential learning model, with one 90-minute class per week. The course includes tennis skill training and social interaction activities that promote cooperation. Compared to conventional physical education courses, this course focuses on enhancing students' collectivism and social responsibility through cooperation and competition in sports.
  Arms: Experimental Group: Tennis Course Based on Experiential Learning Model
Behavioral: Regular Tennis Course — The control group will continue with the regular tennis course, focusing solely on tennis skill development without incorporating the experiential learning model. The course will follow the standard physical education curriculum without additional social interaction activities aimed at enhancing prosocial behavior or cooperation.
  Arms: Control Group: Regular Tennis Course

SUMMARY:
This study adopts a quasi-experimental design and plans to recruit 94 university students from a university in Jiangsu Province, randomly divided into an experimental group and a control group. The experimental group will receive tennis courses based on the experiential learning model, with one 90-minute class each week. The course content will combine tennis skill training and social interaction activities that promote cooperation. The control group will continue with conventional tennis teaching. The study will include baseline testing, teaching intervention, and post-intervention assessment. The main measurement indicators will include prosocial behavior and physical fitness. Prosocial behavior will be evaluated using the PABSS Chinese version questionnaire, which includes aspects such as prosocial behavior toward teammates and opponents, antisocial behavior, and teamwork spirit. Physical fitness will be assessed using the physical fitness test and the CAPL-2 Chinese version questionnaire. Independent samples t-test, paired samples t-test, two-way analysis of variance (ANOVA), and analysis of covariance (ANCOVA) will be used to analyze the differences in prosocial behavior and physical fitness between the experimental and control groups.

ELIGIBILITY:
Inclusion Criteria:

1. Participants are university students aged between 18 and 22 years who are capable of safely participating in physical activities and have no health risks.
2. Students must be able to communicate effectively, understand, and sign the informed consent form.
3. Students must be willing to participate in an 8-week intervention (once a week, 90 minutes per session) and be able to withdraw from the study at any time.
4. Participants must be able to complete all the teaching activities and have no physical or psychological conditions that limit their full participation in physical activities.
5. All participants are from the agreed university in Jiangsu to ensure consistency in the environment and reduce external interference.
6. All participants must agree to follow the study rules and participate in the research.

Exclusion Criteria:

1. Students with physical or psychological health conditions that prevent safe participation in physical activities.
2. Students who are unable to communicate effectively or cannot understand the informed consent form.
3. Students who are unable to attend the full 8-week intervention (once a week, 90 minutes per session).
4. Students who withdraw from the study or do not complete the course during the research period.
5. Students with serious illnesses or health risks will be excluded from the study.
6. Factors such as family socio-economic status, academic performance, or participation in physical activities that could potentially affect the results will be used as exclusion criteria.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2025-09-25 (Actual); Primary Completion 2025-12-12 (Actual); Study Completion 2025-12-12 (Actual)

PRIMARY OUTCOMES:
Prosocial Behavior in University Students After Tennis Course Based On The Experiential Learning Model Intervention | The intervention will last for 8 weeks, with one 90-minute session each week, and outcomes will be measured at the baseline, at the post-intervention stage
  The primary outcome measure is the improvement in prosocial behavior of university students who participated in the tennis course based on the experiential learning model. This will be assessed through the PABSS Chinese version questionnaire , focusing on teamwork, cooperation, social responsibility,
Physical Literacy in University Students After Experiential Learning-Based Tennis Course" | The physical literacy outcomes will be measured at the baseline and post-intervention stage (week 8).
  The primary outcome measure for physical literacy is the improvement in students' overall physical health and fitness after participating in the tennis course based on the experiential learning model. The CAPL-2 Chinese version questionnaire will be used to assess physical literacy based on various aspects of physical health and fitness.

CONTACTS AND LOCATIONS:
Locations (1):
- Yangzhou University, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No